CLINICAL TRIAL: NCT01025765
Title: An Open-label, Multi-center, Randomized Study Comparing the Effects of Oral Hypoglycemic Agents on Viral Kinetics of Chronic Hepatitis C Patients Receiving Pegylated Interferon Alfa 2b Plus Ribavirin
Brief Title: The Effects of Oral Hypoglycemic Agents on Chronic Hepatitis C Patients Receiving Peg-Intron Plus Ribavirin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Schering-Plough (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Jia-Horng Kao, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200905056M
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Pioglitazone; Acarbose; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard care of CHC (No Intervention): From week 5, all the patients will receive Peginterferon alfa-2b (1.5/μg per kg) per week plus Ribavirin 1000-1200 mg/day (≥ 75 kg, 1200 mg; < 75 kg, 1000mg) for 48 weeks.
- Pioglitazone (Experimental): From week 5, all the patients will receive Peginterferon alfa-2b (1.5/μg per kg) per week plus Ribavirin 1000-1200 mg/day (≥ 75 kg, 1200 mg; < 75 kg, 1000mg) for 48 weeks.
  Interventions: Drug: Pioglitazone
- Acarbose (Experimental): From week 5, all the patients will receive Peginterferon alfa-2b (1.5/μg per kg) per week plus Ribavirin 1000-1200 mg/day (≥ 75 kg, 1200 mg; < 75 kg, 1000mg) for 48 weeks.
  Interventions: Drug: Acarbose
- Metformin (Experimental): From week 5, all the patients will receive Peginterferon alfa-2b (1.5/μg per kg) per week plus Ribavirin 1000-1200 mg/day (≥ 75 kg, 1200 mg; < 75 kg, 1000mg) for 48 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone(30mg qd) for 4 weeks of run-in period and 8 weeks of combination treatment with Peginterferon alfa-2b (1.5/μg per kg) per week plus Ribavirin 1000-1200 mg/day (≥ 75 kg, 1200 mg; < 75 kg, 1000mg).
  Arms: Pioglitazone
Drug: Acarbose — Acarbose (50 mg/per meal) for 4 weeks of run-in period and 8 weeks of combination treatment with Peginterferon alfa-2b (1.5/μg per kg) per week plus Ribavirin 1000-1200 mg/day (≥ 75 kg, 1200 mg; < 75 kg, 1000mg).
  Arms: Acarbose
Drug: Metformin — Metformin (500 mg tid) 4 weeks of run-in period and 8 weeks of combination treatment with Peginterferon alfa-2b (1.5/μg per kg) per week plus Ribavirin 1000-1200 mg/day (≥ 75 kg, 1200 mg; < 75 kg, 1000mg). From week 13, all the subjects will receive pegylated interferon alfa plus ribavirin for 40 weeks.
  Arms: Metformin

SUMMARY:
Pegylated interferon in combination with ribavirin is the current standard treatment of chronic hepatitis C virus infection, but is expensive and has several adverse effects. To modify this standard treatment by optimizing its therapeutic effect and decreasing its adverse events are important. Recent studies have identified a close link between metabolic profiles, insulin resistance and Hepatitis C Virus (HCV) infection. Several pilot studies in western world have have found beneficial effects of oral hypoglycemic agents on chronic Hepatitis C (CHC) genotype 1 infected patients. Whether this concept still holds true in Taiwanese people remains unknown.

The objective of this clinical trial is to evaluate the effect of oral hypoglycemic agents (daily for 4 weeks of run-in period and 8 weeks of combination treatment) on CHC genotype 1 infected Taiwanese patients receiving 48 weeks of Peg-IFN plus ribavirin (RBA), and the enrolled subjects will be randomized into 4 treatment groups (including Acarbose, Metformin, Pioglitazone and standard care control groups). During the trial and 24 weeks after the end of treatment, serial serum HCV RNA, alanine aminotransferase (ALT) levels, and other clinical data will be evaluated to determine the therapeutic response and adverse events of the CHC patients.

DETAILED DESCRIPTION:
Pegylated interferon in combination with ribavirin is the current standard treatment of chronic hepatitis C virus infection, but is expensive and has several adverse effects. To modify this standard treatment by optimizing its therapeutic effect and decreasing its adverse events are important.

Recent studies have identified a close link between metabolic profiles, insulin resistance and HCV infection. Chronic hepatitis C (CHC) patients with higher pretreatment HOMA-IR (insulin resistance) index have poor therapeutic response than the ones with lower HOMA-IR index. Thus, it is reasonable to increase the therapeutic response of CHC patients by lowering insulin resistance. Several pilot studies in western world have been conducted to evaluate this concept by adding oral hypoglycemic agents into pegylated interferon plus ribavirin treatment, and have found beneficial effects of oral hypoglycemic agents on CHC genotype 1 infected patients. Whether this concept still holds true in Taiwanese people remains unknown.

To evaluate the effect of oral hypoglycemic agents on CHC genotype 1 infected Taiwanese patients, we design this study and evaluate the virologic, biochemical and histological responses of CHC patients receiving pegylated interferon plus ribavirin treatment, and hope to identify similar beneficial effects of oral hypoglycemic agents in CHC Taiwanese patients.

We plan to enroll about 80 chronic hepatitis C genotype 1 infected patients from the clinics into this study. All patients should have informed consent, not receive any interferon-based therapy or anti-viral medication, abstinence from alcohol beverage for more than 6 months and conformed to the regulations of Bureau of National Health Insurance, Taiwan. All patients will be randomly assigned into 4 different treatment arms. The patients assigned into the first 3 arms will receive one kind of the following oral hypoglycemic agents, such as Acarbose, Metformin, or Pioglitazone for 12 weeks (including 4 weeks of run-in period and 8 weeks of combination treatment with pegylated interferon alfa plus ribavirin). From week 13, all the patients of the first 3 arms will receive pegylated interferon alfa plus ribavirin for 40 weeks. The last arm is the control group; all the patients in the last arm will receive standard pegylated interferon alfa plus ribavirin treatment for 48 weeks. During the trial and 24 weeks after the end of treatment, the serum HCV RNA levels, clinical and biochemical data will be evaluated to determine the therapeutic response and adverse events of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naïve
2. Age old than 18 years old
3. Anti-HCV positive > 6 months
4. Detectable serum quantitative HCV-RNA
5. HCV genotype 1
6. Serum alanine aminotransferase levels above the upper limit of normal with 6 months of enrollment
7. Pre-treatment HOMA-IR ≧ 2.0. (HOMA-IR = fasting insulin (mU/L) x fasting glucose (mg/dL) x 0.05551/22.5)

Exclusion Criteria:

1. Anemia (hemoglobin < 13 gram per deciliter for men and < 12 gram per deciliter for women)
2. Neutropenia (neutrophil count <1,500 per cubic milliliter)
3. Thrombocytopenia (platelet <90,000 per cubic milliliter)
4. Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
5. Chronic alcohol abuse (daily consumption > 20 gram per day in male and >10gram per day in female).
6. Diabetes Mellitus history or under oral hypoglycemic agents therapy Liver cirrhosis
7. Serum creatinine level more than 1.5 times the upper limit of normal Autoimmune liver disease
8. Neoplastic disease
9. An organ transplant
10. Immunosuppressive therapy
11. Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
12. Evidence of drug abuse
13. Unwilling to have contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Response | at the end of 24 weeks post-treatment follow-up

SECONDARY OUTCOMES:
serum ALT normalization, and histologic improvement | at the end of treatment and 24 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Horng Kao, M.D., PhD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Department of Internal Medicine,, Taipei, Taiwan, Taiwan